CLINICAL TRIAL: NCT04182763
Title: A Phase 2 Study of a Vitamin Metabolite for PKAN
Brief Title: CoA-Z in Pantothenate Kinase-associated Neurodegeneration (PKAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Washington State University (Other); Oregon State University (Other); Spoonbill Foundation (Unknown); Spoonbill (Unknown)
Responsible Party: Principal Investigator, Susan J. Hayflick, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00018782; R01HD097328 (NIH)
Record Dates: First submitted 2019-11-24; First posted 2019-12-02 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Pantothenate Kinase-Associated Neurodegeneration
Keywords: Neurodegeneration with Brain Iron Accumulation; NBIA; PKAN
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration

STUDY DESIGN:
Intervention Model Description: An initial 6-month, dose-ranging, parallel-group, randomized, double-blind, placebo-controlled phase is followed by an 18-month, single-dose, open-label phase--these arms met enrollment goals. A direct-to-open-label arm of the study was opened to allow for additional enrollment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking was used for the initial 6-month randomized, double-blind phase, placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- CoA-Z dose 1 (Experimental): 6 months of CoA-Z at the highest assigned dose followed by 18 months of CoA-Z at dose 2
  Interventions: Other: CoA-Z
- CoA-Z dose 2 (Experimental): 6 months of CoA-Z at the medium assigned dose followed by 18 months of CoA-Z at dose 2
  Interventions: Other: CoA-Z
- CoA-Z dose 3 (Experimental): 6 months of CoA-Z at the lowest assigned dose followed by 18 months of CoA-Z at dose 2
  Interventions: Other: CoA-Z
- Placebo (Placebo Comparator): 6 months of placebo, followed by 18 months of CoA-Z at dose 2 (medium dose)
  Interventions: Other: CoA-Z; Other: Placebo
- Open-label arm (Experimental): Up to 24 months of CoA-Z at dose 2
  Interventions: Other: CoA-Z

INTERVENTIONS:
Other: CoA-Z — People with PKAN lack a chemical to process or metabolize a certain vitamin in the brain. CoA-Z is designed to bypass this metabolic defect that causes PKAN.
Other: Placebo — The placebo is a strawberry-flavored syrup that looks and tastes like CoA-Z but has no active CoA-Z in it.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn more about how people with the condition pantothenate kinase-associated neurodegeneration (PKAN) respond to a specialized study product. We are hoping to find out if the study product is safe, what effects-good and bad-the study product causes, and whether the study product changes certain measures of disease in PKAN.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of PKAN confirmed by: a) genetic testing confirming 2 pathogenic or likely pathogenic mutations, or (b) typical findings on exam and brain MR imaging with only one pathogenic mutation +/- a second likely pathogenic or VOUS in PANK2, or (c) typical findings on exam and brain MR imaging with a single likely pathogenic or VOUS in PANK2, or (d) be a symptomatic sibling of a proband subject meeting a, b or c.
* Be between 3 months old and 89 years old.
* Be able to take study product by mouth or feeding tube.
* Be willing and able to complete study procedures / telephone visits / blood draws independently, OR have a caregiver / parent willing and able to assist with these tasks.
* Be enrolled or willing to enroll in the PKANready natural history study (eIRB 10832).
* Be resident in North America (US or Canada) for the duration of the trial.

Exclusion Criteria:

* Have had exposure to a putative PANK2 bypass therapeutic agent in the 30 days prior to screening.
* Be concurrently enrolled in another interventional clinical trial.
* Have concurrent medical or other condition expected to preclude completion of study procedures of confound the assessment of clinical and laboratory measures of safety.

Ages: 3 Months to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penelope Hogarth, M.D., Principal Investigator — Oregon Health and Science University; Susan J Hayflick, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be entered in a stand-alone repository that will allow for future sharing with other researchers. At this time we have not yet determined what IPD are to be shared.
Time Frame: Data will not be available until after September, 2024

REFERENCES:
- See also: Trial information website — http://nbiacure.org/coaz-clinical-trial/

RESULTS

PARTICIPANT FLOW:
Groups:
- CoA-Z Group 1: Double blind CoA-Z 20mg/m^2 (Dose 1) Open label CoA-Z 15mg/m^2 (Dose 2)
- CoA-Z Group 2: Double blind CoA-Z 15mg/m^2 (Dose 2) Open label CoA-Z 15mg/m^2 (Dose 2)
- CoA-Z Group 3: Double blind CoA-Z 5mg/m^2 (Dose 3) Open label CoA-Z 15mg/m^2
- Placebo Group: Double blind CoA-Z Placebo Open label CoA-Z 15mg/m^2
- Open-label arm: Open-label Arm CoA-Z 15mg/m^2
Period: Double-Blind Period, initial 6 months
Arm/Group | CoA-Z Group 1 | CoA-Z Group 2 | CoA-Z Group 3 | Placebo Group | Open-label arm
Started | 15 | 17 | 17 | 16 | 0 (The open-label arm was not divided into 2 phases like the other arms and began in phase 2.)
Completed | 15 | 16 | 17 | 15 | 0
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Period: Open-Label Period, subsequent 18 months
Arm/Group | CoA-Z Group 1 | CoA-Z Group 2 | CoA-Z Group 3 | Placebo Group | Open-label arm
Started | 15 | 16 (Note: the open-label arm was not divided into 2 phases (there was no double-blind phase). Therefore, 12 open-label arm participants are shown as starting their enrollment during phase 2. This means the total enrollment for the study was 77 participants.) | 17 | 15 | 12
Completed | 8 | 9 | 11 | 13 | 10
Not Completed | 7 | 7 | 6 | 2 | 2
Not completed — Death | 3 | 2 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 0 | 1
Not completed — Participation ended early due to shortage of study product (COVID 19 supply chain issue) | 2 | 4 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Note that participants first complete the double-blind period, then crossover to open label, and additional subjects were able to enroll directly into open label. Therefore, the 12 open label participants at baseline are ones who enrolled directly into open label. The others crossed over to open label after the first 6 months and are captured in their original arms.
Groups:
- CoA-Z dose 1: Double blind CoA-Z 20mg/m^2 (Dose 1) Open label CoA-Z 15mg/m^2 (Dose 2)
- CoA-Z dose 2: Double blind CoA-Z 15mg/m^2 (Dose 2) Open label CoA-Z 15mg/m^2 (Dose 2)
- CoA-Z dose 3: Double blind CoA-Z 5mg/m^2 (Dose 3) Open label CoA-Z 15mg/m^2
- Placebo: Double blind CoA-Z Placebo Open label CoA-Z 15mg/m^2
- Open Label: Open-label Arm CoA-Z 15mg/m^2
- Total: Total of all reporting groups
Arm/Group | CoA-Z dose 1 | CoA-Z dose 2 | CoA-Z dose 3 | Placebo | Open Label | Total
Number analyzed (Participants) | 15 | 17 | 17 | 16 | 12 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 11 | 8 | 10 | 44
  Between 18 and 65 years | 8 | 9 | 6 | 8 | 2 | 33
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 5 | 6 | 28
  Male | 10 | 12 | 10 | 11 | 6 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 4 | 5 | 18
  Not Hispanic or Latino | 13 | 12 | 15 | 12 | 7 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1 | 0 | 1 | 3
  Asian | 4 | 0 | 1 | 0 | 0 | 5
  White | 11 | 15 | 14 | 15 | 6 | 61
  Other race | 0 | 1 | 0 | 0 | 4 | 5
  More than one race | 0 | 0 | 1 | 1 | 0 | 2
  Unknown or not reported | 0 | 0 | 0 | 0 | 1 | 1
Type of pantothenate kinase-associated neurodegeneration (PKAN) [Count of Participants; unit: Participants] — Classic disease is defined as onset of motor symptoms by age 5 and loss of ambulation by age 10.
  Atypical PKAN encompasses all participants who are not considered classic.
  Participants
    Classic PKAN | 8 | 9 | 9 | 8 | 4 | 38
    Atypical PKAN | 7 | 8 | 8 | 8 | 8 | 39
Mean number of baseline medications [Mean (Standard Deviation); unit: medications] | 7.7 (6.1) | 6.2 (5.4) | 5.1 (4.0) | 5.6 (4.5) | 2.7 (3.2) | 6.1 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events Assessed Using CTCAE v4.0
Description: Safety will be measured using the number of treatment-emergent adverse events (both AE and SAE) by treatment arm. Counts are adjusted for number of prescription medications at baseline as a measure of baseline disease severity.
Time Frame: 6 months following first dose in double-blind phase
Population: All randomized participants.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Events per person
Arm/Group | CoA-Z dose 1 | CoA-Z dose 2 | CoA-Z dose 3 | Placebo
Number analyzed (Participants) | 15 | 17 | 17 | 16
Events per person | 1.15 [0.78 to 1.52] | 1.38 [0.93 to 1.83] | 1.14 [0.50 to 1.77] | 0.86 [0.55 to 1.16]
Statistical Analysis 1: Comparison: CoA-Z dose 1 vs CoA-Z dose 2 vs CoA-Z dose 3 vs Placebo; Mean counts of events per person were calculated from a negative binomial regression model with categorical coefficients for active dose levels, controlling for the baseline number of prescriptions. A joint test of the null hypothesis that the three regression parameters representing active treatment = 0 was done; Test type: Superiority; p = 0.50, Wald test after neg binomial regression; Chi-squared with 3 d.f

2. Primary Outcome: Number of Treatment-emergent Clinically Significant Laboratory Abnormalities on Complete Blood Count.
Description: Safety will be assessed by measuring the number of treatment-emergent clinically significant laboratory abnormalities on Complete Blood Count. Clinical significance will be determined by Medical Safety Monitor and Clinical Investigators.
Time Frame: 6-month randomized, double-blind, placebo-controlled phase
Measure: Number; unit: Abnormal CBC event
Groups:
- CoA-Z dose 1: 6 months of CoA-Z at the highest assigned dose followed by 18 months at the medium assigned dose.
  CoA-Z: People with PKAN lack a chemical to process or metabolize a certain vitamin in the brain. CoA-Z is designed to bypass this metabolic defect that causes PKAN.
- CoA-Z dose 2: 6 months of CoA-Z at the medium assigned dose followed by 18 months at the medium assigned dose
  CoA-Z: People with PKAN lack a chemical to process or metabolize a certain vitamin in the brain. CoA-Z is designed to bypass this metabolic defect that causes PKAN.
- CoA-Z dose 3: 6 months of CoA-Z at the lowest assigned dose followed by 18 months at the medium assigned dose.
  CoA-Z: People with PKAN lack a chemical to process or metabolize a certain vitamin in the brain. CoA-Z is designed to bypass this metabolic defect that causes PKAN.
- Placebo: 6 months of placebo followed by 18 months of CoA-Z at the medium assigned dose.
  CoA-Z: People with PKAN lack a chemical to process or metabolize a certain vitamin in the brain. CoA-Z is designed to bypass this metabolic defect that causes PKAN.
  Placebo: The placebo is a strawberry-flavored syrup that looks and tastes like CoA-Z but has no active CoA-Z in it.
Arm/Group | CoA-Z dose 1 | CoA-Z dose 2 | CoA-Z dose 3 | Placebo
Number analyzed (Participants) | 15 | 17 | 17 | 16
Abnormal CBC event | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Treatment-emergent Clinically Significant Laboratory Abnormalities on Comprehensive Metabolic Profile.
Description: Safety will be assessed by measuring the number of treatment-emergent clinically significant laboratory abnormalities on Comprehensive Metabolic Profile by collection month. Clinical significance will be determined by Medical Safety Monitor and Clinical Investigators.
Time Frame: 6-month randomized, double-blind, placebo-controlled phase
Measure: Number; unit: Abnormal CMP event
Groups:
- CoA-Z dose 2: 6 months of CoA-Z at the medium assigned dose followed by 18 months at the medium assigned dose.
  CoA-Z: People with PKAN lack a chemical to process or metabolize a certain vitamin in the brain. CoA-Z is designed to bypass this metabolic defect that causes PKAN.
Arm/Group | CoA-Z dose 1 | CoA-Z dose 2 | CoA-Z dose 3 | Placebo
Number analyzed (Participants) | 15 | 17 | 17 | 16
Abnormal CMP event | 1 | 1 | 0 | 0

4. Primary Outcome: Number of Participants Retained in Each Arm.
Description: Tolerability will be assessed by measuring the number of participants retained in each arm over the course of the study.
Time Frame: 6 month randomized, double-blind, placebo-controlled period
Population: All participants who completed Screening, Informed Consent, and enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | CoA-Z dose 1 | CoA-Z dose 2 | CoA-Z dose 3 | Placebo
Number analyzed (Participants) | 15 | 17 | 17 | 16
Participants | 15 | 16 | 17 | 15

5. Primary Outcome: Mean Percent of Study Product Consumed.
Description: Tolerability will be assessed by adherence to the study product regimen arm at each follow-up time point.
Time Frame: 6-month randomized, double-blind, placebo-controlled phase
Population: Population of all subjects who returned partial or complete dosing diaries.
Measure: Mean (Standard Deviation); unit: percent of doses taken
Arm/Group | CoA-Z dose 1 | CoA-Z dose 2 | CoA-Z dose 3 | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 13
percent of doses taken | 98.98 (.014) | 99.25 (.009) | 98.66 (.022) | 96.94 (.048)

6. Secondary Outcome: CoASY mRNA Expression
Description: Average relative CoASY gene expression, measured as the ratio to baseline of 1 / (2^[COASY Ct - 18s Ct]), where Ct = cycle time and 18s is a housekeeping gene. Values >1 reflect higher expression.
Time Frame: Up to 6 months after first dose
Population: All randomized participants
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio to baseline
Arm/Group | CoA-Z dose 1 | CoA-Z dose 2 | CoA-Z dose 3 | Placebo
Number analyzed (Participants) | 15 | 17 | 17 | 16
Ratio to baseline
  1 month +3 days after first dose | 1.31 [1.05 to 1.57] | 1.13 [0.97 to 1.30] | 1.04 [0.86 to 1.22] | 1.07 [0.98 to 1.16]
  6 months after first dose | 1.07 [0.87 to 1.28] | 0.97 [0.77 to 1.16] | 1.02 [0.77 to 1.27] | 0.96 [0.83 to 1.09]
Statistical Analysis 1: Comparison: CoA-Z dose 1 vs CoA-Z dose 2 vs CoA-Z dose 3 vs Placebo; Test that high > med > low > placebo vs the null that all groups are equal at 1 month + 3 days after first dose. Adjusted for PKAN type (classical or atypical), because randomization was stratified on type, and time point; Test type: Superiority; p = 0.105, Linear contrast / test for trend — Two-sided threshold of p<.10; Contrast after mixed-effects GLM with log link, random subject intercept, treatment, PKAN type, and time (1 mo vs 3d)
Statistical Analysis 2: Comparison: CoA-Z dose 1 vs CoA-Z dose 2 vs CoA-Z dose 3 vs Placebo; Test that high > med > low > placebo vs the null that all groups are equal at 6 months after first dose. PKAN type (classical or atypical) was included because randomization was stratified on type. The study hypothesis was that expression levels would not vary significantly at this time point; Test type: Superiority; p = 0.55, Linear contrast / test for trend — Two-sided threshold of p<.10; Contrast after GLM with log link, treatment, and PKAN type

ADVERSE EVENTS:
Time Frame: The 24-month study period for each participant
Description: We included all treatment-emergent adverse events
Groups:
- CoA-Z dose 1 -- double-blind period: Double blind CoA-Z 20mg/m^2 (Dose 1)
- CoA-Z dose 2 -- double-blind period: Double blind CoA-Z 15mg/m^2 (Dose 2)
- CoA-Z dose 3 -- double-blind period: Double blind CoA-Z 5mg/m^2 (Dose 3)
- Placebo -- double-blind period: Double blind CoA-Z Placebo
- CoA-Z dose 1 -- open-label period; CoA-Z dose 2 -- open-label period; CoA-Z dose 3 -- open-label period; Placebo -- open-label period; Open-label period only: Open label CoA-Z 15mg/m^2 (Dose 2)
Arm/Group | CoA-Z dose 1 -- double-blind period | CoA-Z dose 2 -- double-blind period | CoA-Z dose 3 -- double-blind period | Placebo -- double-blind period | CoA-Z dose 1 -- open-label period | CoA-Z dose 2 -- open-label period | CoA-Z dose 3 -- open-label period | Placebo -- open-label period | Open-label period only
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/17 | 0/17 | 0/16 | 3/15 | 2/16 | 2/17 | 0/16 | 1/12
Serious Adverse Events (participants affected / at risk) | 8/15 | 7/17 | 5/17 | 3/16 | 7/15 | 7/16 | 7/17 | 3/16 | 3/12
Other Adverse Events (participants affected / at risk) | 10/15 | 15/17 | 9/17 | 8/16 | 9/15 | 10/16 | 10/17 | 10/16 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoA-Z dose 1 -- double-blind period (N=15) | CoA-Z dose 2 -- double-blind period (N=17) | CoA-Z dose 3 -- double-blind period (N=17) | Placebo -- double-blind period (N=16) | CoA-Z dose 1 -- open-label period (N=15) | CoA-Z dose 2 -- open-label period (N=16) | CoA-Z dose 3 -- open-label period (N=17) | Placebo -- open-label period (N=16) | Open-label period only (N=12)
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive sleep (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
G-tube placement/surgery (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hip dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalization (General disorders) | 2 (6) | 1 (2) | 3 (3) | 0 (0) | 5 (20) | 6 (12) | 6 (10) | 2 (6) | 2 (3)
Mouth injury (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthopedic surgery (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendix rupture (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgery for excessive salivation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Deep brain stimulator placement (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoA-Z dose 1 -- double-blind period (N=15) | CoA-Z dose 2 -- double-blind period (N=17) | CoA-Z dose 3 -- double-blind period (N=17) | Placebo -- double-blind period (N=16) | CoA-Z dose 1 -- open-label period (N=15) | CoA-Z dose 2 -- open-label period (N=16) | CoA-Z dose 3 -- open-label period (N=17) | Placebo -- open-label period (N=16) | Open-label period only (N=12)
Boil (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear tube placement (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated AST (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated LFT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated CK (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
G-tube surgery (outpatient) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Head laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Low platelet count (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MSSA blood infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth sores (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinuplasty (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swimmer's ear (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Whitlow finger (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic dilatation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Barretts esophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Farsighted (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivation, excessive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ADHD (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pressure sore (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial vaginosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne vulgaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Baclofen pump (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth damage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Cauliflower ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematoma drain (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
c. diff infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GERD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone fragment removal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision loss (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysautonomia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anosmia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pes planus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sty (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sialorrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
December 2019, approximately 4 months before the onset of COVID-19 shutdowns. We therefore operated almost entirely during the pandemic, which led to certain challenges. We had to shorten the open-label period for 10 participants due to study product shortage. Additionally, some data presented here are from the 6-month, double-blind, placebo-controlled section of the study, the most important time period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04182763/Prot_SAP_000.pdf